CLINICAL TRIAL: NCT06251492
Title: Radiation and Adebrelimab in Prostate Cancer With Imaging-measurable Disease (RAPID)：a Prospective, Single-arm, Phase II Clinical Study
Brief Title: Radiation and Adebrelimab in Prostate Cancer With Imaging-measurable Disease (RAPID)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, The chair of Department of Urology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPID
Record Dates: First submitted 2024-01-12; First posted 2024-02-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer Metastatic; Castration-resistant Prostate Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Stereotactic body radiotherapy of 8 Gray (Gy) x 3 on targeted metastasis determined by MDT + Adebrelimab 20mg/kg IV every 3 weeks (Q3W) for 2 cycles, then Adebrelimab 20mg/kg IV alone Q3W until progression
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Adebrelimab

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — 8 Gray x 3 for 2 cycles
Drug: Adebrelimab — Adebrelimab 20mg/kg IV Q3W for 2 cycles, then Adebrelimab 20mg/kg IV alone Q3W until progression

SUMMARY:
The aim of this study is to evaluate the efficacy of 2 cycles of combinatory adebrelimab and stereotactic radiotherapy, followed by monotherapy adebrelimab in patients with metastatic castration-resistant prostate cancer. Dr. Yao Zhu from Fudan University Shanghai Cancer Center is the co-leading PI of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male with 18-75 years of age at the time consent form is signed
2. The patient must have histologically or cytologically confirmed prostate adenocarcinoma, which has been determined to be metastatic prostate cancer based on routine imaging assessment (bone scan or CT/MRI);
3. The patient has assessable visceral metastases or soft tissue lesions (outside the pelvis), and the patient should undergo image-guided lesion puncture before medication if considered safe assessed by the PI;
4. Disease progression after treatment with ≥1 androgen-receptor (AR) targeted therapies (such as abiraterone acetate, enzalutamide, apalutamide, darolutamide, etc.);
5. Disease progression after treatment with ≥1 line of taxane-based chemotherapy or intolerant to chemotherapy;
6. The patient shows PSA progression (defined as an increase in PSA levels at least twice consecutively, with an interval of at least one week between assessments, and a PSA value of ≥1 ng/mL at screening), or according to RECIST 1.1 criteria, imaging progression of soft tissue disease with or without PSA progression, or bone lesion progression according to PCWG3 standards: bone scan reveals ≥2 new bone lesions;
7. The patient needs to maintain effective and continuous treatment with luteinizing hormone-releasing hormone analogs (LHRHa) throughout the study treatment, or has undergone orchiectomy; and serum testosterone levels must be maintained at castration level（<50 ng/dL）；
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-2;
9. Expected survival ≥6 months;
10. Normal bone marrow function: absolute neutrophil count ≥1.5×10^9/L; platelets ≥75×10^9/L; hemoglobin ≥90g/L; white blood cell count ≥3.0×10^9/L;
11. Normal liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN); for patients with liver metastases, ALT/AST may be ≤5 times ULN
12. Total bilirubin ≤1.5 times ULN or total bilirubin >1.5 times ULN and direct bilirubin ≤ULN;
13. Normal coagulation function: INR ≤1.5, partial thromboplastin time (APTT) ≤1.5 times ULN, prothrombin time (PT) <ULN+4 seconds;
14. Normal cardiac function: left ventricular ejection fraction (LVEF) ≥50%; QTc <450ms for males, <470ms for females, blood potassium ≥3.5mmol/L;
15. Normal blood pressure: systolic <160mmHg, diastolic <95mmHg; patients with stable blood pressure assessment after appropriate clinical treatment can be enrolled;
16. Normal renal function: serum creatinine ≤1.5 times ULN, and creatinine clearance rate ≥50 mL/min;
17. Researchers consider patients who are capable of ejaculation and are sexually active must agree to take effective contraceptive measures and not donate sperm from the first administration of the study drug to 3 months after the last administration;
18. Able to understand and is willing to sign an informed consent form;
19. Able to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Planning to receive any other antitumor treatments during the study treatment period;
2. Metastatic lesions are limited to bone metastases or include brain metastases;
3. Previous treatment with immune checkpoint inhibitors (including PD-1, PD-L1, CTLA-4 inhibitors, etc.), or antitumor drugs targeting T-cells and activating the immune system;
4. In the past 3 years, having a known other malignancy that is progressing or requiring active treatment. Subjects with skin basal cell carcinoma, skin squamous cell carcinoma, or in situ carcinoma who have received potentially curative treatment may enroll in the study.
5. In the past 2 years, have active autoimmune diseases requiring systemic treatment (such as with disease-modifying drugs, corticosteroids, or immunosuppressive drugs) or active infections (including tuberculosis). Replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for renal or pituitary insufficiency) is not considered systemic treatment.
6. Diagnosed with immunodeficiency or receiving chronic systemic steroid treatment (daily use of more than 10 mg of prednisone or equivalent doses) or any other form of immunosuppressive treatment within 14 days prior to the first dose of the study intervention.
7. Have a history of (non-infectious) pneumonia that required steroid treatment or currently suffering from non-infectious pneumonia.
8. Have received radiation therapy or radionuclide therapy (such as Radium-223) within 28 days prior to the study drug administration; or having been treated with abiraterone within one week prior, with cyproterone acetate within ten days prior, or antiandrogen therapy within two weeks prior.
9. Allergic or intolerant to the active ingredient of PD-L1 monoclonal antibody or any excipient;
10. A clear history of neurological and psychiatric disorders, such as dementia, epilepsy, or a tendency for seizures;
11. In the judgment of the researcher, severe concomitant diseases that pose a serious risk to the subject's safety or affect the subject's completion of the study (such as severe diabetes, thyroid disease, and mental illness, etc.), or the presence of severe and/or unstable medical, psychiatric, or other conditions that affect patient safety or the patient's ability to provide informed consent (including laboratory abnormalities), or any psychological, familial, sociological, or geographical conditions that may affect the study protocol and follow-up plan;
12. The researcher considers the subject unsuitable for participation in the clinical trial for any reason.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | From baseline until progression (up to 24 months)
  DCR (Disease Control Rate) is defined as the proportion of patients with a conﬁrmed complete response (CR) or partial response (PR) of any duration, or stable disease (SD)/non-CR/nonprogressive disease (non-PD) for ≥6 months according to modified Response Evaluation Criteria in Solid Tumours (RECIST1.1) per Prostate Cancer Clinical Trials Working Group (PCWG3) criteria

SECONDARY OUTCOMES:
Objective response rate | From baseline until progression (up to 24 months)
  ORR (objective response rate) is defined as the proportion of patients with a conﬁrmed complete response (CR) or partial response (PR) of any duration according to modified Response Evaluation Criteria in Solid Tumours (RECIST1.1) per Prostate Cancer Clinical Trials Working Group (PCWG3) criteria
Radiographic progression-free survival | From baseline until progression (up to 24 months)
  Defined by radiographic progression by RECIST 1.1 for soft tissue and PCWG3 version 1.1 for bone metastases.
PSA progression-free survival | From baseline until progression (up to 24 months)
  Time to PSA progression as defined by PCWG3 criteria.
PSA response rate | From baseline until progression (up to 24 months)
  PSA response per PCWG3. PSA response is defined as a ≥50% decline in PSA from baseline (measured twice at least 3 weeks apart).
Overall survival | From baseline until progression (up to 24 months)
  Overall survival (OS) is defined as time from start of study treatment to the date of death from any cause. Subjects who are alive will be censored at last follow up date.
Functional Assessment of Quality of life of cancer patients | up to 24 months
  Determined by the FACT-P (Functional Assessment of Cancer Therapy-Prostate) version 4.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fudan University Shanghai Cancer Center Xiamen Branch., Xiamen, Fujian
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No